CLINICAL TRIAL: NCT03180021
Title: Dynamic Imaging of Variation in Lupus Nephritis
Acronym: DIVINE
Status: Completed | Type: Observational
Sponsor: RILITE Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RIL-001
Record Dates: First submitted 2017-04-28; First posted 2017-06-07 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To collect blood and urine samples for future research to identify biomarkers specific to systemic lupus erythematosus and to LN.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Lupus Nephritis
  Interventions: Procedure: MRI
- Patients with IgA Neuropathy
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — This is a multicenter, non-interventional, pilot study. Eligible subjects will have a baseline MRI of the kidney, including anatomical, DWI, BOLD, T1rho, and DCE-MRI, utilizing a macrocyclic gadolinium-based contrast agent (GBCA), followed by planned standard of care (SOC) renal biopsy and clinical laboratory assessments. Additional serum and urine will be collected from subjects at baseline for analysis of research biomarkers. Following the results of the biopsy and clinical laboratory assessments, subjects will be treated for their underlying disease at the discretion of the investigator.
  At 6 months, subjects will return to the clinic for a second MRI, SOC clinical and laboratory evaluation and collection of serum and urine for analysis of research biomarkers.

SUMMARY:
To use a variety of renal imaging modalities, including diffusion weighted imaging (DWI), blood oxygen level dependent (BOLD) imaging, T1rho (T1rho) imaging, and dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) to evaluate the intra-renal blood flow, perfusion, cellularity, fibrosis and atrophy within the kidneys of patients with lupus nephritis (LN) and compare these parameters to renal biopsy findings to determine whether DWI, BOLD, T1rho, and DCE-MRI may provide a set of non-invasive tools to assess renal function and pathology in LN.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent agreeing to all study procedures, before any study- specific procedures are done.
2. Male and female subjects 18 to 65 years of age, inclusive.
3. Subjects currently being evaluated for new or recurrent LN with a SOC kidney biopsy planned OR being evaluated for IgA nephropathy and with a SOC kidney biopsy planned.
4. Patients with LN must meet American College of Rheumatology (ACR) or Systemic Lupus Collaborating Clinics (SLICC) criteria for Systemic Lupus Erythematosus (SLE).
5. Subjects with a life expectancy >6 months.

Exclusion Criteria:

1. Participation in another investigational study during same time period.
2. Contraindication to receiving a GBCA.
3. More than 2 previous lifetime exposures to a GBCA.
4. Any contraindication to MRI, including metal implants, claustrophobia or morbid obesity.
5. Acute or chronic severe renal insufficiency (glomerular filtration rate [GFR] <40 mL per minute per 1.73 m2).
6. Subject requiring dialysis.
7. Presence of pre-existing renal disease unrelated to SLE or IgA nephropathy, respectively.
8. Acute renal insufficiency of any severity caused by the hepato-renal syndrome.
9. Previous or pre-existing nephrogenic systemic fibrosis.
10. History of clinically significant anti-phospholipid syndrome.
11. Chronic liver function impairment, indicated by liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT]) >2-fold upper limit of normal.
12. Platelet count <50,000/μL.
13. Hemoglobin <8.0 g/dL.
14. History of or presence of central nervous system (CNS) disease such as active lupus cerebritis or multiple sclerosis that might compromise blood brain barrier function.
15. Infection that is clinically relevant, particularly hepatitis B virus (HBV), hepatitis C virus (HCV) and/or human immunodeficiency virus (HIV).
16. Pregnant or nursing females, or females not using effective contraception.
17. Inability or unwillingness to return to the research site clinic for study visits at baseline and at 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Lupus Nephritis or IgA neuropathy selected at academic sites listed.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Diffusion Weight Imaging | 7 Months
  Diffusion weighted imaging (DWI) measures ADC values that quantify the combined effects of blood microcirculation and Brownian motion of water molecules within the interstitial space.
Blood Oxygen Level Dependent Imaging | 7 Months
  Blood oxygen level dependent (BOLD) imaging has been widely used to analyze blood flow in various 15 and is the preferred method to detect regional differences in blood flow.
T1rho Imaging | 7 Months
  T1rho (T1rho) imaging is an MRI technique that is sensitive to the presence of macromolecules, such as collagen and proteoglycan 13.
Dynamic Contrast Enhanced Magnetic Resonance Imaging | 7 Months
  Dynamic contrast enhanced (DCE) MRI (DCE-MRI) is an imaging method where T1-weighted MRI scans are acquired dynamically after injection of an MRI contrast agent (e.g., macrocylic gadolinium).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The Regents of the University of Colorado, Aurora, Colorado
  - New York University School of Medicine, New York, New York
  - The Trustees of Columbia University in the City of New York, New York, New York
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No